CLINICAL TRIAL: NCT03282461
Title: A Phase 0 Open Label, Single-center Clinical Trial of ABY-029, an Anti-EGFR Fluorescence Imaging Agent Via Single Intravenous Injection to Subjects With Operable Head and Neck Cancer.
Brief Title: A Microdose Evaluation Study of ABY-029 in Head and Neck Oncology Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Joseph A. Paydarfar, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D17064
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — ABY-029

STUDY DESIGN:
Intervention Model Description: open label
Masking Description: none - open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABY-029 (Experimental): Between 3-9 patients will be administered ABY-029 as a single intravenous injection approximately 1-3 hours prior to surgery.
  Interventions: Drug: ABY-029

INTERVENTIONS:
Drug: ABY-029 — A sample size of 6-12 patients in this open label, single center, clinical trial of ABY-029. Administration will occur as a single intravenous injection to subjects with operable head and neck cancer approximately 1-3 hours prior to surgery.
  Other Names: ABY-029 trifluoroacetate salt; IRDye® 800CW Maleimide labeled Affibody peptide

SUMMARY:
The primary study objective is to determine if microdoses of ABY-029 (up to 6X) lead to detectable signals (defined as signal-to-noise ratio, SNR ≥10, with wide-field iFI) in sampled tissues with an EGFR (epidermal growth factor receptor) pathology score ≥ 1 based on histological staining.

The secondary study objective is to assess ex vivo the specificity of tumor binding in resected specimens by measuring the corresponding molecular uptake and concentrations using histopathology.

DETAILED DESCRIPTION:
The investigators plan to enroll a minimum of 6 and a maximum of 12 adult patients with a diagnosis of operable head and neck cancer in this open label, single center, clinical trial of ABY-029.

Administration of ABY-029 will occur as a single intravenous injection to subjects with operable head and neck cancer approximately 1-3 hours prior to surgery.

Documentation of the tumor with digital photography will be performed at several time points during surgery: pre-resection, at intermediate time points during surgery, and post-resection. White light assessment of the tumor and boundaries will be performed by the surgeon.

Intraoperative optical probe measurements will occur in areas of visible tumor as well as normal appearing tissue. At multiple time points during each surgery and at the discretion of the surgeon, optical probe measurements will be completed with the probe followed by biopsy sampling of the same sites when they are intended for resection. Commonly, these acquisitions will occur at first exposure of the tumor, at the approximate mid-point of tumor resection (when a significant amount of tumor tissue is present in the operative field), at a point nearing but prior to completion of tumor resection (when a small amount of tumor tissue is presumably present), and at the intended completion of tumor resection (when residual tumor may or may not exist). At a data collection time point, optical probe measurements will be performed and archived for analysis and locations may be biopsied when tissue is intended for resection.

Any normal tissue removed as part of surgical procedure will be sampled. Samples may be taken from tissue outside the "antic" tumor volume but resected as part of the procedure along the surgical corridor. All tissue collected will be submitted to pathology for routine processing.

After tissue is removed breadloafed sections will be placed on a fluorescence scanning imager for complete measurement of signal on the exposed surfaces. Pathological analysis for EGFR status will be completed at selected regions around the faces of each breadloaf section.

The protocol is not a safety study since no physiological effects are expected at microdose levels of ABY-029. Rather, doses have been selected to determine if a fluorescence signal can be detected by wide-field imaging technology with a signal-to-noise ratio of 10, which is considered necessary for subsequent assessment of diagnostic performance of ABY-029 as a tumor biomarker sufficient to guide surgical resection in the future. No diagnostic or therapeutic intent is proposed, and study drug administration is not intended to alter the extent of planned tumor resection during the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative diagnosis of head and neck cancer.
2. Tumor judged to be operable based on preoperative imaging studies.
3. Valid informed consent by subject or subject's Legally Authorized Representative.
4. Age ≥ 18 years old.

Exclusion Criteria:

1. Pregnant women or women who are breast feeding.
2. Patients on any experimental anti-EGFR targeted therapies, either investigational or FDA approved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Signal detection | Day of surgery, up to 1 week after surgery
  For each pathology, predictive models of the odds of tumor positivity for biopsies given concentration of ABY-029 will be constructed. Histologically confirmed tumor status from biopsies will be statistically analyzed against the predictive models. The quantitative fluorescence measures will also be assessed for their fit with statistics. The predictive accuracy of the model fit will be summarized through an index.

SECONDARY OUTCOMES:
Correlation of spatial patterns of EGFR expression | within 1 week of surgery
  Regions within the wide-field FI images will be classified as tumor on the basis of their fluorescence signals. Continuous, quantitative optical response data will also be available from the intraoperative probe recordings within the fields-of-view. Two-way classification tables will be examined for agreement between the methods for the "tumor" and "not tumor" categories from an individual patient. Statistical analysis will be used to determine if there is agreement with the region classifications.
  In a second analysis, histopathology from biopsies taken at FI-positive and negative sites will be classified as non-tumor tissue, solid tumor, infiltrating tumor, or indeterminate. The positive predictive values of these locations within the wide-field images will be calculated for each individual. These data will also be analyzed for sensitivity and specificity of the fluorescence image signatures relative to the reference standard (histopathology).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Paydarfar, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT03282461/ICF_000.pdf